CLINICAL TRIAL: NCT06444555
Title: Nutritional Needs and Food Supplement Intake of Adolescent Girls in Burkina Faso and Ethiopia
Brief Title: Adolescent Nutrition in Girls in Burkina Faso and Ethiopia
Acronym: Adonut
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Addis Continental Institute of Public Health (Other); Institut de Recherche en Sciences de la Sante, Burkina Faso (Other Government); Bill and Melinda Gates Foundation (Other); AfricSanté, Burkina Faso (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ONZ-2024-0038
Record Dates: First submitted 2024-05-21; First posted 2024-06-05 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Nutrition Deficiency Due to Insufficient Food

STUDY DESIGN:
Intervention Model Description: 200 adolescent girls will be enrolled in Ethiopia and 200 adolescent girls will be enrolled in Burkina Faso.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Balanced Energy Protein Supplement (Experimental): Fortified lipid-based nutrient supplement
  Interventions: Dietary Supplement: BEP supplement
- Multiple Micronutrient Supplement (Active Comparator): The United Nations International Multiple Micronutrient Antenatal Preparation (UNIMMAP).
  Interventions: Dietary Supplement: Multiple Micronutrient supplement

INTERVENTIONS:
Dietary Supplement: BEP supplement — The BEP supplement used in Burkina Faso is a fortified medium-quantity lipid-based nutrient supplement called Plumpy'Doz. The product is a peanut and milk-based ready-to-use nutritional formulation produced by Nutriset. A peanut-based BEP formulation with a trademark Plumpy'Sup produced by Hilina Enriched Foods PLC will be used in Ethiopia.
  Other Names: Balanced energy protein supplement
  Arms: Balanced Energy Protein Supplement
Dietary Supplement: Multiple Micronutrient supplement — The MMN formulation is based on the United Nations International Multiple Micronutrient Antenatal Preparation (UNIMMAP). The formulation contains 15 minerals and vitamins and is administered as a tablet.
  Other Names: UNIMAPP
  Arms: Multiple Micronutrient Supplement

SUMMARY:
Adolescents' diets are key to breaking the intergenerational cycle of malnutrition. This study will guide policies and programs on the adequacy, acceptability, and feasibility of implementing balanced energy protein and multiple micronutrient supplementations to fill nutrient gaps in adolescent girls. Using a trial, the study will assess dietary intake and nutrient gaps, acceptability of balanced energy protein and multiple micronutrient supplementations. In addition to the trial, the study will the assess willingness to pay for the supplements and the most effective delivery platform and model to reach vulnerable adolescent girls. The most effective delivery platform and model to reach vulnerable adolescent girls cost-effectively will also be assessed through interviews with (inter)national experts, producers, and the donor community.

DETAILED DESCRIPTION:
In low- and middle-income countries, it is estimated that each year, 21 million adolescent girls become mothers. Infants of adolescent mothers are at increased risk of delivering babies preterm, with low birth weight or length. Targeting nutrition interventions to improve adolescent girls' diet and nutrition is crucial to breaking the intergenerational cycle of poor growth and development. There is a specific need to assess how a balanced energy protein (BEP) and multiple micronutrient (MMN) supplement interventions can be tailored to adolescent girls and women of reproductive age.

This study aims to assess the adequacy, acceptability, and feasibility of implementing nutritional supplementations to fill nutrient gaps in adolescent girls in resource-limited settings. A trial will specifically:

1. assess the short-term acceptability of BEP and MMN supplements
2. assess how nutrition supplements increase nutrient adequacy of diets adolescent girls in resources-limited settings;

Using a qualitative component, the study explores the food agency of adolescents and the most effective delivery platform to reach vulnerable adolescent girls cost-effectively. The overall aim is to guide policies and programs on new formulations of nutritional supplements for adolescent girls in resource-limited settings.

ELIGIBILITY:
Eligibility criteria are all based on self-reported information

Inclusion criteria:

* Non-pregnant and non-lactating women
* Without any known chronic illness or acute illness affecting appetite
* Permanent residents of the study area

Exclusion criteria:

* Being allergic to peanuts
* Eating disorders or dietary restrictions

Ages: 15 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Only females are recruited.
Enrollment: 400 (Actual)
Dates: Start 2024-05-28 (Actual); Primary Completion 2024-07-05 (Actual); Study Completion 2024-07-05 (Actual)

PRIMARY OUTCOMES:
Acceptability of the supplement | Day 8 (after 7 days of consumption)
  Acceptability to the nutritional supplements, as measured using a 9-item scale (1 "Dislike extremely" up to 9 "Like extremely")
Nutritional adequacy | Day 8 (after 7 days of consumption)
  Mean nutrient adequacy ratio of adolescent diets, using 24 h recall

SECONDARY OUTCOMES:
Willingness to pay for the supplement | Day 8 (after 7 days of consumption)
  Mean household head's willingness to pay values elicited through their bids
Reported consumption of the supplement | Day 8 (average of 7-day intervention)
  Percent of the recommended nutritional supplement consumed during the intervention period, self-reported
Substitution of food and nutrient intake | Day 8 (after 7 days of consumption)
  Substitution of food and nutrition intake at group level, using 24 h recall
Nutrient intake | Day 8 (after 7 days of consumption)
  Mean energy, macronutrient and micronutrient intake between the BEP and MMN group, using 24 h recall

CONTACTS AND LOCATIONS:
Overall Officials: Yemane Berhane, Prof, Principal Investigator — Addis Continental Institute of Public Health; Firehiwot Workneh, dr., Study Director — Addis Continental Institute of Public Health; Moustapha Drabo, Dr, Study Director — University Ghent; Carl Lachat, Prof, Study Chair — University Ghent; Laeticia Céline Toé, MD, Principal Investigator — Institute de Recherche en Sciences de la Santé, Bobo Dioulasso; Hans De Steur, Prof, Principal Investigator — University Ghent; Alemayehu Alemayehu, Dr, Principal Investigator — University Ghent
Locations (2):
- Agence de Formation, de Recherche et d'Expertise en Santé pour l'Afrique (AFRICSanté), Bobo-Dioulasso, Burkina Faso
- Addis Continental Institute of Public Health, Addis Ababa, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes
The data will be transferred to the donor in a pseudo-anonymised way. After preparing a data-sharing agreement, the investigators will also share food intake data with the Food and Agriculture Organization and World Health Organization (FAO/WHO) of the United Nations Global Individual Food Consumption Data Tool. All research output generated by the project is open access as part of the Grant Agreement with the funder. Given the personal nature of the data, individual data will only be shared after a data transfer agreement with third parties. The informed consent form mentions that data can be shared outside the study team.
Time Frame: Individual participant data will be shared after data cleaning and quality checks are completed. All study other study materials will be shared after the finalization of the data collection.
Access Criteria: Personal data will only be shared under a data sharing agreement, subject to approval by the relevant authorities. The transfer will only be performed in the public interest, which means that it will increase knowledge and insight to society's direct or indirect benefit.